CLINICAL TRIAL: NCT06174779
Title: A Multicenter, Randomized, Double-blind, Phase 3 Study to Evaluate Efficacy and Safety of HM11260C in Adult Obesity Patients Without Diabetes Mellitus
Brief Title: A Study to Evaluate Efficacy and Safety of HM11260C in Adult Obesity Patients Without Diabetes Mellitus
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM-EXC-301
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HM11260C (Experimental): Weekly administration by subcutaneous injection
  Interventions: Drug: HM11260C
- Placebo (Placebo Comparator): Weekly administration by subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HM11260C — Test drug
  Arms: HM11260C
Drug: Placebo — Placebo drug
  Arms: Placebo

SUMMARY:
A multicenter, randomized, double-blind, phase 3 study to evaluate efficacy and safety of HM11260C in adult obesity patients without diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

1. Patients with following criteria :

   * BMI ≥ 30 kg/m2 or
   * 27 kg/m2 ≤ BMI < 30 kg/m2 with more than one risk factors or comorbidities(hypertension, dyslipidemia, sleep apnea, cardiocerebrovascular disease)
2. A person who have failed at least once to weight control using diet and exercise therapy before screening visit.

Exclusion Criteria:

1. A person whose weight change exceeds 5kg within 3 months prior to screening visit.
2. Diabetes mellitus (Type 1, type 2, etc.) or HbA1c ≥ 6.5 %.
3. Administration of hypoglycemic agents.
4. Administration of medicines inducing weight gain.
5. Prader-Willi Syndrome or MC4R deficiency.
6. Cushing's Syndrome.
7. Administration of medicines for weight management.
8. A person who has a history of surgery(including device-based therapy) related to obesity or who has a plan during the clinical trial period.
9. Administration of Steroids for the systemic use.
10. Clinically significant gastric emptying abnormalities.
11. History(including family history) of medullary thyroid carcinoma or multiple endocrine adenomatosis.
12. History of acute or chronic pancreatitis.
13. A person who has the following clinical laboratory test results :

    * TSH < 0.4 mIU/L or TSH > 6 mIU/L
    * Calcitonin > 100 ng/L
    * Amylase or Lipase > 3 x UNL
14. Severe liver disease (AST or AST > 3 x UNL or Total bilirubin > 1.5 x UNL).
15. Severe renal disease ( eGFR < 30mL/min/1.73m 2 ).
16. QTc > 450 ms.
17. Answered 'yes' to question 4 or 5 of the suicidal ideation domain in C-SSRS or history of suicide attempt.
18. PHQ-9 ≥ 15 or history of depression, anxiety, and other severe Mental illness.
19. History of alcohol addiction or drug abuse.
20. History of malignant tumors.
21. History of severe heart disease or severe neurovascular disease.
22. Hypersensitivity to investigational products or multi-drug allergy.
23. Positive to pregnancy test, nursing mother, intention on pregnancy.
24. Considered by investigator as not appropriate to participate in the clinical study with other reason.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
The percent change of body weight from baseline | baseline, 40 weeks
The proportion of subjects achieving body weight loss ≥ 5% from baseline | baseline, 40 weeks

SECONDARY OUTCOMES:
The percent change of body weight from baseline | baseline, 24 weeks, 64 weeks
The proportion of subjects achieving body weight loss ≥ 5% from baseline | baseline, 24 weeks, 64 weeks
The proportion of subjects achieving body weight loss ≥ 10% from baseline | baseline, 24 weeks, 40 weeks, 64 weeks
Change of body weight from baseline | baseline, 24 weeks, 40 weeks, 64 weeks
Change of BMI from baseline | baseline, 24 weeks, 40 weeks, 64 weeks
Change of waist circumference from baseline | baseline, 24 weeks, 40 weeks, 64 weeks
Change of glucose metabolism parameters from baseline | baseline, 24 weeks, 40 weeks, 64 weeks
The percentage change of lipid profile parameters from baseline | baseline, 24 weeks, 40 weeks, 64 weeks
Change of blood pressure from baseline | baseline, 24 weeks, 40 weeks, 64 weeks
Change of IWQoL-Lite-CT(Physical function domain) from baseline | baseline, 24 weeks, 40 weeks, 64 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kangbuk samsung hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No